CLINICAL TRIAL: NCT05753072
Title: Value and Impact of a Stakeholder-operationalised Carer Support Nurse Role and Feasibility of a Future Wider Implementation Study
Brief Title: Value and Impact of a Carer Support Nurse
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: Health Education England, Wessex (Other); NIHR Applied Research Collaboration - East of England (Unknown); UEA Health & Social Care Partners (Unknown); University of Hertfordshire (Other); London South Bank University (Other); Norfolk & Waveney ICB (Unknown)
Responsible Party: Sponsor
Other Study IDs: R211343
Record Dates: First submitted 2023-02-08; First posted 2023-03-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-02

CONDITIONS: Not Condition Specific
Keywords: unpaid carers; family carers; specialist nurse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Carer Support Nurse — Specialist community nursing role to support unpaid family/carers with complex health-related support needs or unresolved health-related support needs that cannot be met by their usual health care team

SUMMARY:
Families and friends play a crucial role supporting people they care for as their unpaid carers. However, they are not always well prepared for this, and it can damage their own health and wellbeing. This can impact their ability to keep 'caring'. Carers often lack time to look after themselves, putting their own needs last. These needs tend to be hidden until crises. Carers need support to (1) look after their own health and wellbeing and (2) boost their skills and confidence to care. Healthcare policy says this should happen, but healthcare professionals can find this difficult alongside supporting the patient.

To address this, we have worked with carers, health and social care professionals, voluntary organisations and national leaders in carer support, to develop a new Carer Support Nurse role. This role is designed to help carers who have their own needs, or who need extra support for their caring role, that cannot be met by their usual healthcare team. The nurse will also work with other healthcare providers to raise their awareness of carer needs and how to support them.

The Carer Support Nurse is now in post. This study explores the role's value and impact by analysing data on (1) what the nurse does, and (2) the views of carers, patients, health and social care professionals, voluntary organisations, and the nurse themself. This will involve collecting data from (1) the nurse (through a weekly diary and monthly interviews), (2) carers who have had contact with the nurse (through a survey and interviews), (3) patients these carers support (through interviews), and (4) health and social care professionals and voluntary organisations (through interviews and focus groups). It will also develop recommendations for whether, and how, the role could be introduced more widely, and the design of a future multi-site study.

DETAILED DESCRIPTION:
Five-task study using qualitative and quantitative data to answer its research questions. Sample sizes are indicators rather than target sample sizes.

TASK 1) Carer Support Nurse role data capture:

The Carer Support Nurse (CSN) will receive a recruitment pack comprising an invitation letter, participant information sheet, and with reply by email. The CSN job description informed applicants of the research being conducted alongside the role, and it was discussed at interview. The CSN will therefore expect to receive the recruitment pack and will have an opportunity to ask further questions before informed consent is taken.

Once consented, the CSN will complete a very brief templated Weekly Reflective Diary [Gabbay, 2003] (what was done, what worked, what didn't) and CSNAT-I Activity Template (anonymised group-level data on carer needs identified and types of actions taken: no names/identifiers included). Monthly data-generating meetings (informed by the data collected weekly) will monitor how the role is working and identify/address any emerging barriers to the role. Additionally, an adapted version of a tool designed to capture the activities the nurse is carrying out within the role will be used (the Cassandra tool [https://www.apollonursingresource.com/showing-how-i-spend-my-time/cassandra-app/]) and costs. Data collected through these monthly meetings will include:

* referral sources (including repeat referrals)
* CSN's use of time (e.g., working hours, activities with carers, activities not directly with carers)
* delivery of five Evidence-based Design Principles for the role, or whether these had to be modified
* types of actions taken in response to carers' needs
* potential impacts (costs/benefits) on the CSN, carers, patients, or other services.

This will provide evidence on the value and cost of the role and help commissioners understand what activities are undertaken to achieve the role's outcomes and how complex the CSN's work is. The monthly meetings will not be audio-recorded but notes will be taken onto a template (method used successfully previously). The activities the nurse carries out within the role (e.g., types of interventions, for whom, where) will be compared with an established dataset of activities usually carried out by other specialist nursing roles [Punshon et al, 2019], to inform how the role is working.

Each month anonymised group-level data will be provided by the site (aggregated data at a group or system level, rather than for individual carers e.g., number of carers seen by the CSN, number of repeat contacts). This will inform the design of a future multi-site study e.g., population description, carer needs identified, actions taken to meet needs, costs, capacity, cost-per-carer.

Task 1 will run in parallel with Task 2 below.

TASK 2) Carer outcomes and experiences of carers and patients:

Once the CSN is established in the post with a working caseload (estimated three months into post), carers who have had contact with the nurse will be invited to participate in the study. It is estimated that the nurse will see about 120 carers during the planned 6-month data collection period for this task. Carer baseline and outcome data will be collected from adult carers who have contact with the nurse through a baseline and follow up postal survey, and interviews with a sub-sample of carers. Patients will also be invited to be interviewed.

The CSN will provide carers who fit the study inclusion/exclusion criteria with a recruitment pack for the study. It will include an invitation letter, participant information sheet, consent form and baseline Carer Postal Survey Booklet. The participant information sheet will include contact details for the research team should the carer have any questions. The invitation letter and participant information sheet will invite carers to complete the baseline survey, a follow up survey, and potentially be contacted for interview. Those carers willing to receive a follow-up survey, and/or potentially be contacted for interview, will provide their contact details on a reply form. Carers may opt not to complete the follow-up survey but still to take part in the interview. The recruitment pack was developed with our Carer PPI group.

The Baseline Carer Postal Survey Booklet, reviewed by our Carer PPI group, includes six items:

* Item 1: Preparedness for Caregiving Scale (8 items) [Archbold et al, 1990]
* Item 2: Warwick-Edinburgh Mental Wellbeing Scale (7 items) [Stewart-Brown, 2009; https://warwick.ac.uk/fac/sci/med/research/platform/wemwbs/about/]
* Item 3: EQ-5D-5L (6 item health status questionnaire) [Feng et al, 2021; https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/]
* Item 4: resource use questions (in last 6 weeks) e.g., primary care, secondary care, social care, respite care
* Item 5: contact with the CSN (as could occur) and planned appointments
* Item 6: background questions: age, sex, ethnic group, number of people carer is supporting, living situation (i.e., with patient(s)/distance from patient(s)), relationship to patient(s), patient's(s') primary diagnosis, caregiving hours, employment status, funding status (receipt of funded care) The Follow-up Carer Postal Survey Booklet will be sent (to consenters) approximately six weeks from the carer's first contact with the CSN. It will include items 1-5 only (not 6).

Interviews with a sub-sample of carers (and the patients they support) who have received the CSN intervention will explore their experiences of the CSN, ideally within two weeks of their main CSN contact (about 12 carers will be sought in order to provide enough data - known as "information power" [Malterud et al, 2016]). Purposive sampling will seek as much variation in this sub-sample as possible in relation to carer sex, age and ethnic group. Data on the timing of interviews (in relation to the carers' contacts with the nurse) will be collected to inform the design of a future multi-site study. Carers who earlier agreed to be contacted for interview, and who meet the purposive sampling criteria, will be contacted by letter, email, or phone (depending on their indicated preference) to invite them to be interviewed.

These carers will also be asked if the research team can send them an additional recruitment pack for the patient they support, inviting the patient to also be interviewed (separately). If the contact with the carer about the interview is by letter, then the patient recruitment pack will be included with it to optionally share with the patient; if the contact with the carer is by email or phone, the patient recruitment pack will be sent to the carer to share with the patient if the carer agrees. The patient recruitment pack will include an invitation letter, participant information sheet, with reply-options by email, post, or at the end or the start of the carer interview (if they live in the same household).

Carers and patients will be able to ask any questions before informed consent is taken (online, by email or by post). The topic-guided interviews will be conducted online or by phone. They will be audio-recorded (with permission), then transcribed by a professional transcription company. The research team will then anonymise them and analyse the anonymised transcripts using a method called framework analysis [Ritchie et al, 2003]. The carer interview topic guide will cover their caring role, support they may have had before contact with the CSN, their contact with the CSN, and what was helpful or unhelpful about it. The patient interview topic guide will explore whether patients felt the CSN was helpful, or if anything was unhelpful, and any impact it has had on them as the patient. The interviews will also help inform the design of a future multi-site study.

TASK 3) Experiences and impacts from the viewpoint of the CSN and colleagues from different sectors:

End of study interviews with the CSN and their line manager (interviewed separately) and focus groups with key colleagues from different sectors (health, social care and the voluntary sector) will explore:

* the role (experiences of delivering it, or working alongside it)
* role activity (e.g., activities with carers, activities not directly with carers, activities with colleagues)
* whether the CSN delivered the five Evidence-based Design Principles or whether they were modified and how (and the impact of this)
* perceived impacts (positive/negative)
* mechanisms of action (how the role worked)
* barriers, enablers and strategies influencing implementation of the role
* learnings for the design of a future multi-site study.

The line manager interview and cross-sector colleague focus groups will additionally explore:

• impacts on own (or team members') awareness of, attitudes to, and engagement with carers, subsequent to the CSN starting in post.

For Task 3, the CSN will already have been recruited at Task 1. The CSN's line manager will be invited to take part in Task 3 via an emailed recruitment pack from the study team. The line manager is already in contact with the research team. The recruitment pack will include an invitation letter and participant information sheet, with reply by email (directly back to the study team). They will have an opportunity to ask any questions before informed consent is taken (in person or online depending on interview mode). The interviews will be topic guided and audio-recorded (with permission), and will either be conducted in person, online or by phone.

The focus groups (two in total to enable people to take part, but they will only attend one of them) will involve health, social and voluntary sector working partners (up to nine participants in total, across the two groups). These key cross-sector colleagues will be identified first from the CSN's role activity in the preceding months, and secondly through other stakeholders consulted during study work-up (from across health settings, social care, voluntary sector, and HealthWatch) if needed to ensure representation of each sector. These cross-sector colleagues will be invited to participate via an emailed recruitment pack (an invitation letter, participant information sheet) with reply by email. They will have an opportunity to ask any questions before informed consent is taken (online or by email). The focus groups will be topic guided and audio-recorded (with permission) and conducted online.

The interview and focus group audio-recordings will be transcribed, anonymised, then analysed using framework analysis [Ritchie et al, 2003].

TASK 4) Establishing mechanisms of action and effect and recommendations:

The core team, our Carer PPI group and Project Advisory Group will bring together the findings of Task 1-3 to explore whether and how the role worked. The findings will also inform any suggestions for improving the CSN role going forward. We will then work together to develop recommendations on whether and how to keep the role going and introduce it elsewhere. This will also inform the design of a future multi-site study.

FUTURE WORK

If the CSN role shows promise, funding will be sought to further develop and evaluate the role in a future multi-site study informed by the feasibility data gathered.

ELIGIBILITY:
Inclusion Criteria:

* Adult unpaid carers who have been referred to, or who have contacted (self-referral), the Carer Support Nurse

Exclusion Criteria:

* Unable to understand or communicate in English
* Serious mental health problem
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unpaid/family carers with complex health-related support needs or unresolved health-related support needs that cannot be met by their usual health care team
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Carer Preparedness for Caregiving | 6 weeks
  Preparedness for Caregiving Scale

SECONDARY OUTCOMES:
Carer wellbeing | 6 weeks
  Warwick-Edinburgh Mental Wellbeing Scale
Health-related quality of life | 6 weeks
  EQ-5D-5L
Carer resource use | 6 weeks
  Carer resource use questions e.g., primary care, secondary care, social care, respite care

CONTACTS AND LOCATIONS:
Overall Officials: Morag Farquhar, PhD, Principal Investigator — University of East Anglia (UEA)
Locations (1):
- East Coast Community Health Care, Great Yarmouth, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabbay J, le May A, Jefferson H, et al. A Case Study of Knowledge Management in Multiagency Consumer-Informed 'Communities of Practice': Implications for Evidence-Based Policy Development in Health and Social Services. Health. 2003;7(3):283-310.
- [Background] https://www.apollonursingresource.com/showing-how-i-spend-my-time/cassandra-app/
- [Background] Punshon G, Sopala J, Hannan G, Roberts M, Vernon K, Pearce A, Leary A. Modeling the Multiple Sclerosis Specialist Nurse Workforce by Determination of Optimum Caseloads in the United Kingdom. Int J MS Care. 2021 Jan-Feb;23(1):1-7. doi: 10.7224/1537-2073.2019-058. Epub 2020 Jan 13. PMID 33658899
- [Background] Archbold PG, Stewart BJ, Greenlick MR, Harvath T. Mutuality and preparedness as predictors of caregiver role strain. Res Nurs Health. 1990 Dec;13(6):375-84. doi: 10.1002/nur.4770130605. PMID 2270302
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] https://warwick.ac.uk/fac/sci/med/research/platform/wemwbs/about/
- [Background] https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Malterud K, Siersma VD, Guassora AD. Sample Size in Qualitative Interview Studies: Guided by Information Power. Qual Health Res. 2016 Nov;26(13):1753-1760. doi: 10.1177/1049732315617444. Epub 2016 Jul 10. PMID 26613970
- [Background] Ritchie J et al. Qualitative Research Practice. Sage 2003
- See also: Carer Support Nurse pilot — https://arc-eoe.nihr.ac.uk/research-implementation/research-themes/palliative-and-end-life-care/carer-support-nurse-pilot